CLINICAL TRIAL: NCT00002969
Title: Phase II Trial of Paclitaxel by 96-Hour Infusion in Stage IIIB and IV Bronchioloalveolar Carcinoma (BAC)
Brief Title: S9714: Paclitaxel in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065476; S9714 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy with paclitaxel in treating patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess survival, progression-free survival and response rate of patients with bronchioloalveolar carcinoma receiving paclitaxel. II. Evaluate toxic effects of paclitaxel in 96 hour continuous infusion patients.

OUTLINE: Patients receive 6 cycles of paclitaxel by IV continuous infusion over 96 hours. Before cycle 4, restaging is performed. If disease progression is witnessed, patients are removed from the study. If a stable, partial, or complete response is observed, patients receive the total of 6 cycles. Three weeks after the last cycle, final restaging is performed. Patients are followed every 3 months while on treatment and every 6 months thereafter, unless more frequent follow-up is clinically recommended.

PROJECTED ACCRUAL: 50 patients will be enrolled. The accrual rate is estimated at 25 per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven Stage IIIB or IV bronchioloalveolar non-small cell lung carcinoma -incompletely resected or unresectable -tumors may be multifocal or diffuse -measurable or evaluable disease required No prior brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: SWOG 0-2 Life Expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than institutional upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine no greater than institutional ULN OR creatinine clearance at least 50 mL/min Other: Not pregnant or nursing Effective contraceptive method used while on study No prior malignancies allowed, except: basal or squamous cell skin cancer in situ cervical cancer Stage I or II cancer which is in remission Any cancer from which patients have been disease free for 5 years

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior biologic therapy for lung cancer Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiation therapy (including palliative radiotherapy) Surgery: Prior surgery is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1997-05; Primary Completion 2004-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph B. Vance, MD, Study Chair — University of Mississippi Cancer Clinic
Locations (85):
- United States (85):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Beckman Research Institute, City of Hope, Duarte, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Medical Center, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - CCOP - Central Illinois, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Hospital - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Ozarks Regional, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Hospital Tumor Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- [Background] Gandara DR, West H, Chansky K, Davies AM, Lau DH, Crowley J, Gumerlock PH, Hirsch FR, Franklin WA. Bronchioloalveolar carcinoma: a model for investigating the biology of epidermal growth factor receptor inhibition. Clin Cancer Res. 2004 Jun 15;10(12 Pt 2):4205s-4209s. doi: 10.1158/1078-0432.CCR-040012. PMID 15217959
- [Result] West HL, Crowley JJ, Vance RB, Franklin WA, Livingston RB, Dakhil SR, Giguere JK, Rivkin SE, Kraut M, Chansky K, Gandara DR; Southwest Oncology Group. Advanced bronchioloalveolar carcinoma: a phase II trial of paclitaxel by 96-hour infusion (SWOG 9714): a Southwest Oncology Group study. Ann Oncol. 2005 Jul;16(7):1076-80. doi: 10.1093/annonc/mdi215. Epub 2005 Apr 28. PMID 15860488
- [Result] Franklin WA, Gumerlock PH, Crowley J, et al.: EGFR, HER2 and ERB-B pathway activation in bronchioloalveolar carcinoma (BAC): analysis of SWOG 9417 and lung SPORE tissue samples. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2493, 2003.
- [Result] Vance RB, Crowly JJ, Livingston RB, et al.: A phase II Southwest Oncology Group trial (S9714) utilizing paclitaxel by 96-hour infusion in stage IIIb and IV bronchioloalveolar carcinoma of the lung (BAC). [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1340, 336a, 2001.